CLINICAL TRIAL: NCT05081154
Title: An In-Clinic Confinement Study to Assess Nicotine Uptake From P10 Nicotine Pouches
Brief Title: CSD201002: Study to Assess Nicotine Uptake From P10 Nicotine Pouches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD201002
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Product usage order A B G C F D E (Experimental): Subjects will use each of the 7 products (A B G C F D E) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order B C A D G E F (Experimental): Subjects will use each of the 7 products (B C A D G E F) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order C D B E A F G (Experimental): Subjects will use each of the 7 products (C D B E A F G) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order D E C F B G A (Experimental): Subjects will use each of the 7 products (D E C F B G A) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order E F D G C A B (Experimental): Subjects will use each of the 7 products (E F D G C A B) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order F G E A D B C (Experimental): Subjects will use each of the 7 products (F G E A D B C) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order G A F B E C D (Experimental): Subjects will use each of the 7 products (G A F B E C D) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order E D F C G B A (Experimental): Subjects will use each of the 7 products (E D F C G B A) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order F E G D A C B (Experimental): Subjects will use each of the 7 products (F E G D A C B) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order G F A E B D C (Experimental): Subjects will use each of the 7 products (G F A E B D C) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order A G B F C E D (Experimental): Subjects will use each of the 7 products (A G B F C E D) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order B A C G D F E (Experimental): Subjects will use each of the 7 products (B A C G D F E) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order C B D A E G F (Experimental): Subjects will use each of the 7 products (C B D A E G F) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Product usage order D C E B F A G (Experimental): Subjects will use each of the 7 products (D C E B F A G) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G

INTERVENTIONS:
Other: Product A — P1012915, a nicotine pouch with 8 mg nicotine
Other: Product B — P1013018, a nicotine pouch with 10 mg nicotine
Other: Product C — P1013015, a nicotine pouch with 8 mg nicotine
Other: Product D — P1012815, a nicotine pouch with 8 mg nicotine
Other: Product E — P1013315, a nicotine pouch with 8 mg nicotine
Other: Product F — P1013115, a nicotine pouch with 8 mg nicotine
Other: Product G — P1013215, a nicotine pouch with 8 mg nicotine

SUMMARY:
This study is a single-center, open-label, randomized, 7-way crossover study designed to evaluate plasma nicotine pharmacokinetics (PK) parameters following use of the study investigational products (IPs) in a confinement setting by generally healthy combustible cigarette (CC) smokers.

DETAILED DESCRIPTION:
This study is designed to evaluate plasma nicotine PK parameters following the use of nicotine pouches (hereinafter referred to as Velo Pouch IPs) in cigarette smokers and smokers who also use smokeless tobacco (SST) [e.g., snus, moist snuff]. At least one-third of the study population will include smokers who also use ST.

Potential subjects may complete a pre-screening telephone interview. They will complete a Screening Visit to assess their eligibility within 45 days prior to enrollment, randomization and confinement.

Following the Screening Visit, eligible subjects will be scheduled for a Day 1 check-in visit to complete procedures to confirm eligibility. Eligible subjects will be enrolled and begin confinement at the clinical site for 8 days and 7 nights. Subjects will participate in separate Test Sessions for plasma nicotine PK assessment, one for each IP. The IP for each Test Session will be determined based on a randomly assigned IP presentation schedule (14 product sequence) generated using a Williams Design. Each Test Session will last for approximately 4 hours following the start of the IP use, and will include collection of plasma samples for PK assessments prior to, during and following IP use and completion of the Overall Product Liking questionnaire. Subjects will use their randomized study IP one day before the respective test session to familiarize themselves with the IP.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy males or females, 21 to 60 years of age, inclusive, at the time of consent.
3. Smokes combustible, filtered, non-menthol or menthol cigarettes, 83 mm to 100 mm in length as primary source of tobacco.
4. Smokers who also use ST products (e.g., moist snuff, snus), and have used ST within 30 days prior to screening will be enrolled.
5. Smokes an average of at least 10 cigarettes per day (CPD) and inhale the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the PI.
6. Agrees to smoke the same Usual Brand (UB) cigarette throughout the study period. The UB cigarette is defined as the reported cigarette brand and style currently smoked most frequently by the subject.
7. Expired breath carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at Screening and at check-in Day 1.
8. Positive urine cotinine test at Screening.
9. Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes" (Heatherton et al., 1991).
10. Willing to use the UB cigarette and Velo Pouch IPs during the study period.
11. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to the start of each of seven Test Sessions.
12. Females must be willing to use a form of contraception acceptable to the PI from the time of signing the informed consent until End-of-Study.

    Examples of acceptable means of birth control are, but not limited to: a) Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy, bilateral salpingectomy); b) physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide; c) non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs (e.g., Mirena or Kyleena); d) vasectomized partner; and e) post-menopausal and not on hormone replacement therapy.
13. Agrees to an in-clinic confinement of 8 days (7 nights).

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
4. History or presence of bleeding or clotting disorders.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
6. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at Screening and at check-in Day 1.
7. Weight of ≤ 110 pounds.
8. Hemoglobin level is < 12.5 g/dL for females or <13.0 g/dL for males at Screening.
9. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
10. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or check-in Day 1.
11. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
12. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
13. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or self-reports a previous quit attempt within (≤) 30 days prior to the signing the informed consent.
14. Any use of daily aspirin (≥ 325 mg/day) or any use of other anticoagulants.
15. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
16. Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent and between Screening and check-in Day 1.
17. Plasma donation within (≤) 7 days prior to signing the informed consent and between Screening and check-in Day 1.
18. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
19. Participation in another clinical trial within (≤) 30 days prior to signing the informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the informed consent in the current study.
20. Drinks more than 21 servings of alcoholic beverages per week
21. Has a positive alcohol result at Screening or check-in Day 1.
22. Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
AUC nic 0-240 | 0 to 240 minutes
  Baseline-adjusted area under the plasma nicotine concentration-versus-time curve from time zero to 240 minutes after the start of IP use
Cmax | 240 minutes
  Maximum baseline-adjusted plasma concentration of nicotine

CONTACTS AND LOCATIONS:
Overall Officials: Milly Kanobe, PhD, Study Director — RAIS
Locations (1):
- AMR Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kanobe MN, Powell CY, Patrudu M, Baxter SA, Tapia MA, Darnell J, Prevette K, Gibson AG, Ayoku SA, Campbell L, Coffield JW, Keyser BM, Ganesh BS, Gale N, Jordan KG. Randomized crossover clinical studies to assess abuse liability and nicotine pharmacokinetics of Velo Oral Nicotine pouches. Front Pharmacol. 2025 Mar 13;16:1547073. doi: 10.3389/fphar.2025.1547073. eCollection 2025. PMID 40183092